CLINICAL TRIAL: NCT06829147
Title: Development and Validation of a Deep Learning Model for Diagnosing Lymph Node Metastasis in Nasopharyngeal Carcinoma Using Histologic Whole Slide Images and Time-dependent Magnetic Resonance Images
Brief Title: A Deep Learning Model for Diagnosing Lymph Node Metastasis in Nasopharyngeal Carcinoma(NPC)
Acronym: NPC
Status: Recruiting | Type: Observational
Sponsor: Sun Yat-sen University (Other)
Collaborators: First People's Hospital of Foshan (Other); Affiliated Cancer Hospital & Institute of Guangzhou Medical University (Other); Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other)
Responsible Party: Principal Investigator, Pu-Yun OuYang, Associate Chief Physician, Sun Yat-sen University
Other Study IDs: B2024-769-01
Record Dates: First submitted 2025-02-08; First posted 2025-02-17 (Actual); Last update posted 2025-02-17 (Actual); Status verified 2025-02

CONDITIONS: Nasopharyngeal Cancinoma (NPC); Lymph Node Metastasis
Keywords: Nasopharyngeal carcinoma; Cervical lymph node metastasis; MRI; pathology; Artificial Intelligence Diagnostic Model
MeSH Terms: conditions — Lymphatic Metastasis; Nasopharyngeal Carcinoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Prospective Validation Cohort: Prospective patient enrollment to validate the diagnostic efficacy of the AI model

SUMMARY:
(I) AI Model for Diagnosing Lymph Node Metastasis We developed an AI model to help diagnose whether a single lymph node in nasopharyngeal cancer has spread. The model uses MRI images of the lymph node and the area around it. It includes: 1.Automatically identifying the lymph nodes and the primary tumor. 2.Analyzing MRI images of the lymph node and surrounding area. 3.Using MRI scans before and after chemotherapy to track changes in the lymph node.

(II) AI Model for Predicting Lymph Node Metastasis We created an AI model that predicts whether a lymph node in a specific area has cancer. This model uses a combination of the primary tumor's pathology and MRI images of both the tumor and lymph node. It also tracks changes in the lymph node over time. The model includes: 1.Analyzing the tumor's pathology to identify specific lymphatic structures. 2.Using MRI scans to predict the likelihood of metastasis in a single lymph node. 3.Examining MRI scans before and after chemotherapy to help determine if the lymph node has metastasized.

(III) Verifying and Analyzing the Benefits of the AI Model We are testing the AI model to see how well it works and its potential benefits, including: 1.Checking if the AI can correct past diagnoses of recurrent lymph nodes in nasopharyngeal cancer, which could help guide treatment plans for radiotherapy. 2.Testing the model using biopsy results from head and neck cancer patients to see if it can accurately detect negative lymph nodes. 3.Running clinical trials to test the AI model's safety and effectiveness in guiding radiation treatment for upper neck and single lymph node areas in nasopharyngeal cancer. 4.Analyzing the economic benefits of using the AI model in radiation treatment for nasopharyngeal cancer.

DETAILED DESCRIPTION:
(I) AI Model for Assisting Diagnosis of Lymph Node Metastasis in Nasopharyngeal Carcinoma Based on MRI Features of the Lymph Node and Surrounding 3mm Area.

An AI model is developed to assist in diagnosing whether a single lymph node in nasopharyngeal carcinoma has metastasized, based on the MRI features of the lymph node itself and its surrounding 3mm area. Specifically, the model includes: 1.Automatic segmentation of the lymph node and primary lesion using a semi-supervised AI model. 2.Construction of a single dual-view AI model based on baseline MRI features of the lymph node itself and its surrounding 3mm area. 3.Development of a dual-time series dual-view AI model based on MRI features of the lymph nodes before and after induction chemotherapy.

(II) Multimodal AI Model for Predicting Lymph Node Metastasis. A multimodal AI model is constructed to predict metastasis of a single station lymph node and diagnose lymph node metastasis "from surface to point." This is based on pathological features of the nasopharyngeal primary lesion, MRI images, lymph node location, and other factors. Specifically, the model includes: 1.Construction of an AI model based on H&E stained digital pathology of the primary lesion to extract features of the tertiary lymphatic structure. 2.Development of a multimodal AI model integrating pathological features of the nasopharyngeal primary lesion and baseline MRI images of both the primary lesion and lymph node to predict the probability of lymph node metastasis in a single station. 3.Construction of a single or dual-time series multimodal AI model using the probability of lymph node metastasis and baseline MRI or two MRI scans before and after induction chemotherapy to diagnose whether a single lymph node in the station has metastasized.

(III) Verification and Economic Benefit Analysis of AI Models. The AI models are subjected to thorough verification and economic benefit analysis. Specifically, the process includes: 1.Retrospective correction of historical diagnoses of in situ recurrent lymph nodes in nasopharyngeal carcinoma patients using the AI model to verify its potential benefits in guiding prescription doses for single lymph node radiotherapy. 2.Validation of the AI model using pathological results from lymph node dissection in head and neck squamous cell carcinoma patients to assess the detection rate of clinically diagnosed negative lymph nodes. 3.Prospective clinical trials to evaluate the effectiveness and safety of the AI model in guiding prescription doses for upper neck radiotherapy and single lymph node radiotherapy in nasopharyngeal carcinoma patients. 4.Economic benefit analysis to illustrate the economic value of the AI model in guiding upper neck radiotherapy for nasopharyngeal carcinoma.

ELIGIBILITY:
Inclusion Criteria:

1. The primary lesion was pathologically confirmed as nasopharyngeal carcinoma (WHO classification is I, II and III);
2. MRI scan was performed at the initial diagnosis (before anti-tumor treatment), and transverse and coronal MRI images before treatment were available, including T1-weighted, T2-weighted and T1-enhanced scanning sequences.
3. PET/CT scan was performed at the initial diagnosis (before anti-tumor treatment)
4. When MRI and PET/CT were inconsistent in judging the benign or malignant nature of lymph nodes, the patient agreed to undergo cervical lymph node puncture and pathological examination.

Exclusion Criteria:

1. The patient has undergone cervical lymph node radiotherapy for any reason
2. Combined with other malignant tumors

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with pathologically confirmed nasopharyngeal carcinoma
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2024-11-19 (Actual); Primary Completion 2026-09-01 (Estimated); Study Completion 2026-09-01 (Estimated)

PRIMARY OUTCOMES:
AUC | through study completion, an average of 2 year
  AUC (Area Under the Curve) refers to the area under a performance curve, typically the ROC (Receiver Operating Characteristic) curve or PR (Precision-Recall) curve, that is used to evaluate the performance of a classification model. It is a single scalar value that provides an aggregate measure of a model's ability to distinguish between classes (e.g., positive and negative samples).

SECONDARY OUTCOMES:
Sensitivity and Specificity | through study completion, an average of 2 year
  Sensitivity and Specificity are fundamental metrics used to evaluate the performance of a classification model, especially in medical diagnostics, machine learning, and statistics. These metrics are used to measure how well a model can correctly identify positive and negative cases.

OTHER OUTCOMES:
Positive Predictive Value (PPV) and Negative Predictive Value (NPV) | through study completion, an average of 2 year
  Positive Predictive Value (PPV) and Negative Predictive Value (NPV) are performance metrics used to evaluate the reliability of a model's predictions, particularly in binary classification tasks. These metrics focus on the accuracy of the model's positive and negative predictions.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Radiation Oncology, Sun Yat-sen University Cancer Center, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) might not be shared due to concerns about patient privacy, ethical considerations, or institutional policies. Restrictions may also arise from data protection regulations, confidentiality agreements, or the potential risk of re-identification. Additionally, if the data includes sensitive medical information, sharing may require special approvals or de-identification processes that are not feasible.

REFERENCES:
- [Background] Liu Y, Lai F, Lin B, Gu Y, Chen L, Chen G, Xiao H, Luo S, Pang Y, Xiong D, Li B, Peng S, Lv W, Alexander EK, Xiao H. Deep learning to predict cervical lymph node metastasis from intraoperative frozen section of tumour in papillary thyroid carcinoma: a multicentre diagnostic study. EClinicalMedicine. 2023 May 18;60:102007. doi: 10.1016/j.eclinm.2023.102007. eCollection 2023 Jun. PMID 37251623
- [Background] Wessels F, Schmitt M, Krieghoff-Henning E, Jutzi T, Worst TS, Waldbillig F, Neuberger M, Maron RC, Steeg M, Gaiser T, Hekler A, Utikal JS, von Kalle C, Frohling S, Michel MS, Nuhn P, Brinker TJ. Deep learning approach to predict lymph node metastasis directly from primary tumour histology in prostate cancer. BJU Int. 2021 Sep;128(3):352-360. doi: 10.1111/bju.15386. Epub 2021 May 5. PMID 33706408
- [Background] Chen C, Zhang Y, Wu X, Shen J. The role of tertiary lymphoid structure and B cells in nasopharyngeal carcinoma: Based on bioinformatics and experimental verification. Transl Oncol. 2024 Mar;41:101885. doi: 10.1016/j.tranon.2024.101885. Epub 2024 Jan 31. PMID 38295746
- [Background] Wibawa MS, Zhou JY, Wang R, Huang YY, Zhan Z, Chen X, Lv X, Young LS, Rajpoot N. AI-Based Risk Score from Tumour-Infiltrating Lymphocyte Predicts Locoregional-Free Survival in Nasopharyngeal Carcinoma. Cancers (Basel). 2023 Dec 10;15(24):5789. doi: 10.3390/cancers15245789. PMID 38136336
- [Background] Haggstrom I, Leithner D, Alven J, Campanella G, Abusamra M, Zhang H, Chhabra S, Beer L, Haug A, Salles G, Raderer M, Staber PB, Becker A, Hricak H, Fuchs TJ, Schoder H, Mayerhoefer ME. Deep learning for [18F]fluorodeoxyglucose-PET-CT classification in patients with lymphoma: a dual-centre retrospective analysis. Lancet Digit Health. 2024 Feb;6(2):e114-e125. doi: 10.1016/S2589-7500(23)00203-0. Epub 2023 Dec 21. PMID 38135556
- [Background] Zhong Y, Cai C, Chen T, Gui H, Chen C, Deng J, Yang M, Yu B, Song Y, Wang T, Chen Y, Shi H, Xie D, Chen C, She Y. PET/CT-based deep learning grading signature to optimize surgical decisions for clinical stage I invasive lung adenocarcinoma and biologic basis under its prediction: a multicenter study. Eur J Nucl Med Mol Imaging. 2024 Jan;51(2):521-534. doi: 10.1007/s00259-023-06434-7. Epub 2023 Sep 19. PMID 37725128
- [Background] Lee JO, Ahn SS, Choi KS, Lee J, Jang J, Park JH, Hwang I, Park CK, Park SH, Chung JW, Choi SH. Added prognostic value of 3D deep learning-derived features from preoperative MRI for adult-type diffuse gliomas. Neuro Oncol. 2024 Mar 4;26(3):571-580. doi: 10.1093/neuonc/noad202. PMID 37855826
- [Background] OuYang PY, Zhang BY, Guo JG, Liu JN, Li J, Peng QH, Yang SS, He Y, Liu ZQ, Zhao YN, Li A, Wu YS, Hu XF, Chen C, Han F, You KY, Xie FY. Deep learning-based precise prediction and early detection of radiation-induced temporal lobe injury for nasopharyngeal carcinoma. EClinicalMedicine. 2023 Apr 4;58:101930. doi: 10.1016/j.eclinm.2023.101930. eCollection 2023 Apr. PMID 37090437
- [Background] Jiang C, Gong B, Gao H, Zhang T, Li Z, Wang J, Zhang L. Correlation analysis of neck node levels in 960 cases of Nasopharyngeal carcinoma (NPC). Radiother Oncol. 2021 Aug;161:23-28. doi: 10.1016/j.radonc.2021.05.020. Epub 2021 May 25. PMID 34044063
- [Background] Zhu GL, Zhang XM, Yang KB, Tang LL, Ma J. Metastatic patterns of level II-V cervical lymph nodes assessed per vertebral levels in nasopharyngeal carcinoma. Radiother Oncol. 2023 Feb;179:109447. doi: 10.1016/j.radonc.2022.109447. Epub 2022 Dec 19. PMID 36549338
- [Background] Meng Z, Li P, Yang D, Huang H, Dong H, Qin Y, Bin Y, Li R, Wang S, Chen X, Kang M. The feasibility of level Ib-sparing intensity-modulated radiation therapy in patients with nasopharyngeal carcinoma and high-risk factors classified based on the International Guideline. Radiother Oncol. 2024 Feb;191:110027. doi: 10.1016/j.radonc.2023.110027. Epub 2023 Nov 24. PMID 38008418
- [Background] Yao JJ, Qi ZY, Liu ZG, Jiang GM, Xu XW, Chen SY, Zhu FT, Zhang WJ, Lawrence WR, Ma J, Zhou GQ, Sun Y. Clinical features and survival outcomes between ascending and descending types of nasopharyngeal carcinoma in the intensity-modulated radiotherapy era: A big-data intelligence platform-based analysis. Radiother Oncol. 2019 Aug;137:137-144. doi: 10.1016/j.radonc.2019.04.025. Epub 2019 May 15. PMID 31102988
- [Background] Fang J, Wang J, Li A, Yan Y, Liu H, Li J, Yang H, Hou Y, Yang X, Yang M, Liu J. Parameterized Gompertz-Guided Morphological AutoEncoder for Predicting Pulmonary Nodule Growth. IEEE Trans Med Imaging. 2023 Dec;42(12):3602-3613. doi: 10.1109/TMI.2023.3297209. Epub 2023 Nov 30. PMID 37471191
- [Background] Venkadesh KV, Aleef TA, Scholten ET, Saghir Z, Silva M, Sverzellati N, Pastorino U, van Ginneken B, Prokop M, Jacobs C. Prior CT Improves Deep Learning for Malignancy Risk Estimation of Screening-detected Pulmonary Nodules. Radiology. 2023 Aug;308(2):e223308. doi: 10.1148/radiol.223308. PMID 37526548
- [Background] Kolk MZH, Ruiperez-Campillo S, Alvarez-Florez L, Deb B, Bekkers EJ, Allaart CP, Van Der Lingen ACJ, Clopton P, Isgum I, Wilde AAM, Knops RE, Narayan SM, Tjong FVY. Dynamic prediction of malignant ventricular arrhythmias using neural networks in patients with an implantable cardioverter-defibrillator. EBioMedicine. 2024 Jan;99:104937. doi: 10.1016/j.ebiom.2023.104937. Epub 2023 Dec 19. PMID 38118401
- [Background] Zhang Y, Chen L, Hu GQ, Zhang N, Zhu XD, Yang KY, Jin F, Shi M, Chen YP, Hu WH, Cheng ZB, Wang SY, Tian Y, Wang XC, Sun Y, Li JG, Li WF, Li YH, Mao YP, Zhou GQ, Sun R, Liu X, Guo R, Long GX, Liang SQ, Li L, Huang J, Long JH, Zang J, Liu QD, Zou L, Su QF, Zheng BM, Xiao Y, Guo Y, Han F, Mo HY, Lv JW, Du XJ, Xu C, Liu N, Li YQ, Xie FY, Sun Y, Ma J, Tang LL. Final Overall Survival Analysis of Gemcitabine and Cisplatin Induction Chemotherapy in Nasopharyngeal Carcinoma: A Multicenter, Randomized Phase III Trial. J Clin Oncol. 2022 Aug 1;40(22):2420-2425. doi: 10.1200/JCO.22.00327. Epub 2022 Jun 16. PMID 35709465
- [Background] Sher DJ, Moon DH, Vo D, Wang J, Chen L, Dohopolski M, Hughes R, Sumer BD, Ahn C, Avkshtol V. Efficacy and Quality-of-Life Following Involved Nodal Radiotherapy for Head and Neck Squamous Cell Carcinoma: The INRT-AIR Phase II Clinical Trial. Clin Cancer Res. 2023 Sep 1;29(17):3284-3291. doi: 10.1158/1078-0432.CCR-23-0334. PMID 37363993
- [Background] Kann BH, Likitlersuang J, Bontempi D, Ye Z, Aneja S, Bakst R, Kelly HR, Juliano AF, Payabvash S, Guenette JP, Uppaluri R, Margalit DN, Schoenfeld JD, Tishler RB, Haddad R, Aerts HJWL, Garcia JJ, Flamand Y, Subramaniam RM, Burtness BA, Ferris RL. Screening for extranodal extension in HPV-associated oropharyngeal carcinoma: evaluation of a CT-based deep learning algorithm in patient data from a multicentre, randomised de-escalation trial. Lancet Digit Health. 2023 Jun;5(6):e360-e369. doi: 10.1016/S2589-7500(23)00046-8. Epub 2023 Apr 21. PMID 37087370
- [Background] Wang W, Liang H, Zhang Z, Xu C, Wei D, Li W, Qian Y, Zhang L, Liu J, Lei D. Comparing three-dimensional and two-dimensional deep-learning, radiomics, and fusion models for predicting occult lymph node metastasis in laryngeal squamous cell carcinoma based on CT imaging: a multicentre, retrospective, diagnostic study. EClinicalMedicine. 2024 Jan 3;67:102385. doi: 10.1016/j.eclinm.2023.102385. eCollection 2024 Jan. PMID 38261897
- [Background] OuYang PY, He Y, Guo JG, Liu JN, Wang ZL, Li A, Li J, Yang SS, Zhang X, Fan W, Wu YS, Liu ZQ, Zhang BY, Zhao YN, Gao MY, Zhang WJ, Xie CM, Xie FY. Artificial intelligence aided precise detection of local recurrence on MRI for nasopharyngeal carcinoma: a multicenter cohort study. EClinicalMedicine. 2023 Aug 30;63:102202. doi: 10.1016/j.eclinm.2023.102202. eCollection 2023 Sep. PMID 37680944
- [Background] Shen G, Xiao W, Han F, Fan W, Lin XP, Lu L, Zheng L, Yue N, Haffty B, Zhao C, Deng X. Advantage of PET/CT in Target Delineation of MRI-negative Cervical Lymph Nodes In Intensity-Modulated Radiation Therapy Planning for Nasopharyngeal Carcinoma. J Cancer. 2017 Nov 6;8(19):4117-4123. doi: 10.7150/jca.21582. eCollection 2017. PMID 29187888
- [Background] van den Brekel MW, Stel HV, Castelijns JA, Nauta JJ, van der Waal I, Valk J, Meyer CJ, Snow GB. Cervical lymph node metastasis: assessment of radiologic criteria. Radiology. 1990 Nov;177(2):379-84. doi: 10.1148/radiology.177.2.2217772.
- [Background] Yang SS, Wu YS, Pang YJ, Xiao SM, Zhang BY, Liu ZQ, Chen EN, Zhang X, OuYang PY, Xie FY. Development and validation of radiologic scores for guiding individualized induction chemotherapy in T3N1M0 nasopharyngeal carcinoma. Eur Radiol. 2022 Jun;32(6):3649-3660. doi: 10.1007/s00330-021-08460-1. Epub 2022 Jan 6. PMID 34989842
- [Background] Yang SS, Wu YS, Chen WC, Zhang J, Xiao SM, Zhang BY, Liu ZQ, Chen EN, Zhang X, OuYang PY, Xie FY. Benefit of [18F]-FDG PET/CT for treatment-naive nasopharyngeal carcinoma. Eur J Nucl Med Mol Imaging. 2022 Feb;49(3):980-991. doi: 10.1007/s00259-021-05540-8. Epub 2021 Sep 1. PMID 34468782